CLINICAL TRIAL: NCT05153629
Title: Noninvasive Electrical Stimulator as an Adjunct for Pain Control After Ureteroscopic Stone Management
Brief Title: Noninvasive Electrical Stimulator as a Pain Control Treatment Post-ureteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Simon Conti, Clinical Assistant Professor, Urology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-62416
Record Dates: First submitted 2021-11-28; First posted 2021-12-10 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Kidney Stone; Ureteral Calculi; Nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi; Nephrolithiasis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard care (No Intervention): Participants will follow standard care until the ureteral stent is removed
- TENS device (Experimental): Participants will use the TENS device until the ureteral stent is removed
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — TENS device used four times a day for 60 minutes each time
  Arms: TENS device

SUMMARY:
The investigators will assess the use of Transcutaneous Neurostimulation (TENS), a pharmacological alternative, for treatment of ureteral stent pain post-ureteroscopy. The primary aim for the investigators is to determine if use of a TENS unit will reduce post-operative pain and nausea associated with the ureteral stent. Secondary aim will be to assess if it can help minimize narcotic use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing standard of care ureteroscopy and laser lithotripsy for urinary stone disease
* Patients receiving a stent following their ureteroscopy and laser lithotripsy

Exclusion Criteria:

* Children
* Pregnant patients
* Patients unable to answer pain questionnaire
* Patients undergoing PCNL
* Patients being treated for Urologic malignancy with ureteroscopy
* Patients who require long term or chronic ureteral stent management
* Patient with implantable stimulators
* Patient with epilepsy
* Patients undergoing laser lithotripsy without stent placement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Conti, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 participant signed consent; 30 were randomized
Groups:
- TENS Device: Participants use the TENS device (four times a day for 60 minutes each time) until the ureteral stent is removed
- Standard Care: Participants follow standard care until the ureteral stent is removed
Period: Overall Study
Arm/Group | TENS Device | Standard Care
Started | 17 | 13
Completed | 17 | 11
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | TENS Device | Standard Care | Total
Number analyzed (Participants) | 17 | 11 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.94 (14.38) | 63.09 (15.79) | 56.92 (15.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 16 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 0 | 5
  African American | 1 | 0 | 1
  White | 8 | 9 | 17
  Other | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 11 | 28
Surgical Laterality [Count of Participants; unit: Participants]
  Right | 6 | 5 | 11
  Left | 11 | 6 | 17
Stone Location [Count of Participants; unit: Participants]
  Ureteral | 8 | 3 | 11
  Renal | 8 | 5 | 13
  Both | 1 | 3 | 4
Stent Length in cm [Count of Participants; unit: Participants]
  20 | 3 | 1 | 4
  22 | 4 | 0 | 4
  24 | 5 | 5 | 10
  26 | 5 | 4 | 9
  28 | 0 | 1 | 1
Concomitant Anxiety/Depression [Count of Participants; unit: Participants] | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Pain on 11-point Visual Analog Score Scale (VAS)
Description: Cumulative average pain score using an 11-point VAS. The VAS is a validated tool widely used to assess pain intensity. Possible score ranges:
  * Scale for back pain: 0 (no pain) - 10 (worst pain)
  * Abdominal/Groin Pain: 0 (no pain) - 10 (worst pain)
  * Pain Frequency: 0 (not at all) - 10 (All day or night long)
  * Nausea intensity: 0 (No nausea) - 10 (Worst possible nausea)
Time Frame: Assessed daily until removal of stent, approximately 3-10 days after placement
Population: Participants who completed the protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS Device | Standard Care
Number analyzed (Participants) | 17 | 11
score on a scale
  Back Pain | 3.52 (3.08) | 3.42 (2.85)
  Abdominal/Groin Pain | 4.44 (2.59) | 4.02 (2.44)
  Pain Frequency | 4.70 (2.33) | 5.22 (2.28)
  Nausea Intensity | 1.18 (1.63) | 1.98 (2.01)
Statistical Analysis 1: Comparison: TENS Device vs Standard Care; Analysis of back pain; Test type: Other; p = 0.93, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 2: Comparison: TENS Device vs Standard Care; Analysis of abdominal/groin pain; Test type: Other; p = 0.76, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 3: Comparison: TENS Device vs Standard Care; Analysis of pain frequency; Test type: Other; p = 0.56, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 4: Comparison: TENS Device vs Standard Care; Analysis of nausea intensity; Test type: Other; p = 0.26, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant

2. Primary Outcome: Difference in Pain on 11-point Visual Analog Score Scale (VAS)
Description: Cumulative average difference in pain score using an 11-point VAS. The VAS is a validated tool widely used to assess pain intensity. Possible score ranges:
  * Scale for back pain: 0 (no pain) - 10 (worst pain)
  * Abdominal/Groin Pain: 0 (no pain) - 10 (worst pain)
  * Pain Frequency: 0 (not at all) - 10 (All day or night long)
  * Nausea intensity: 0 (No nausea) - 10 (Worst possible nausea)
Time Frame: Assessed daily until removal of stent, approximately 3-10 days after placement
Population: Participants who completed the protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS Device | Standard Care
Number analyzed (Participants) | 17 | 11
score on a scale
  Back Pain | -3.94 (6.59) | -6.09 (10.29)
  Abdominal/Groin Pain | -4.88 (9.55) | -8.54 (7.74)
  Pain Frequency | -5.64 (7.52) | -8.63 (9.50)
  Nausea Intensity | -1.05 (4.97) | -4.09 (7.58)
Statistical Analysis 1: Comparison: TENS Device vs Standard Care; Analysis of difference in back pain; Test type: Other; p = 0.55, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 2: Comparison: TENS Device vs Standard Care; Analysis of difference in abdominal/groin pain; Test type: Other; p = 0.28, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 3: Comparison: TENS Device vs Standard Care; Analysis of difference in pain frequency; Test type: Other; p = 0.39, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 4: Comparison: TENS Device vs Standard Care; Analysis of difference in nausea intensity; Test type: Other; p = 0.26, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant

3. Secondary Outcome: Total Opioid Consumption
Description: Consumption in morphine milligram equivalents (MME), based on patient-self-report in Daily Symptom Questionnaire.
Time Frame: Until stent removal (up to 10 days)
Population: Participants who completed the protocol
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | TENS Device | Standard Care
Number analyzed (Participants) | 17 | 11
MME | 31.73 (66.08) | 17.27 (28.21)
Statistical Analysis 1: Comparison: TENS Device vs Standard Care; Test type: Other; p = 0.50, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant

4. Secondary Outcome: Difference in Total Opioid Consumption
Description: Consumption (in MME), based on patient-self-report in Daily Symptom Questionnaire.
Time Frame: Until stent removal (up to 10 days)
Population: Participants who completed the protocol
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | TENS Device | Standard Care
Number analyzed (Participants) | 17 | 11
MME | -5.03 (25.64) | 2.72 (31.23)
Statistical Analysis 1: Comparison: TENS Device vs Standard Care; Test type: Other; p = 0.50, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant

5. Secondary Outcome: Ureteral Stent Discomfort Test (USDT) Scale Score
Description: Overall score scale:0 to 61 points; subdomain scales: urinary symptoms: 0 to 30; pain: 0 to 6: daily life: 0 to 5; sexual life: 0 to 5; medical care/analgesic use: 0 to 10; and overall quality of life: 0 to 5. Subscale scores are totaled to calculate the overall score. Higher scores correspond to more severe symptoms for the overall score and all subscale scores.
Time Frame: Assessed at removal of stent, approximately 3-10 days after placement
Population: Participants who completed the USDT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS Device | Standard Care
Number analyzed (Participants) | 13 | 10
score on a scale
  Overall score | 30.23 (6.48) | 29.30 (11.02)
  Urinary symptoms | 16.92 (4.89) | 16.00 (7.20)
  Pain | 3.15 (1.52) | 2.70 (1.57)
  Daily life | 2.54 (1.39) | 3.10 (1.91)
  Sexual life | 0.08 (0.28) | 0.50 (1.58)
  Medical care/analgesic use | 4.23 (2.17) | 3.60 (2.07)
  Overall Quality of Life | 3.31 (1.32) | 3.40 (1.51)
Statistical Analysis 1: Comparison: TENS Device vs Standard Care; Analysis of overall USDT score; Test type: Other; p = 0.80, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 2: Comparison: TENS Device vs Standard Care; Analysis of urinary symptoms; Test type: Other; p = 0.72, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 3: Comparison: TENS Device vs Standard Care; Analysis of pain; Test type: Other; p = 0.45, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 4: Comparison: TENS Device vs Standard Care; Analysis of daily life; Test type: Other; p = 0.42, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 5: Comparison: TENS Device vs Standard Care; Analysis of sexual life; Test type: Other; p = 0.36, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 6: Comparison: TENS Device vs Standard Care; Analysis of medical care/analgesic use; Test type: Other; p = 0.49, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant
Statistical Analysis 7: Comparison: TENS Device vs Standard Care; Analysis of overall quality of life; Test type: Other; p = 0.88, t-test, 2 sided — A p-value less than the a priori threshold of 0.05 is considered statistically significant

6. Secondary Outcome: Patient Satisfaction Survey
Description: Participants were asked if they would prefer using TENS over pain medication during a pain episode, and whether they would consider using TENS over pain medication in the future. This outcome was assessed only in participants who were randomized to the TENS device group.
Time Frame: End of study (day 3 to 10)
Population: Participants who received the TENS device and completed the survey questions
Measure: Count of Participants; unit: Participants
Arm/Group | TENS Device
Number analyzed (Participants) | 13
Participants
  Preferred TENS device over medication | 9
  Would use TENS device in the future | 12

ADVERSE EVENTS:
Time Frame: Up to 10 days
Arm/Group | TENS Device | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 0/17 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT05153629/Prot_SAP_000.pdf